CLINICAL TRIAL: NCT05857930
Title: A Randomized, Placebo-Controlled, Double-Blind, Multicenter, Phase 2 Study to Assess the Efficacy and Safety of Daily OM-85 Treatment vs. Placebo Given in Children Aged 6 Months to 5 Years With Recurrent Wheezing
Brief Title: A Study to Assess the Efficacy and Safety of Daily OM-85 in Young Children With Recurrent Wheezing
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OM Pharma SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BV-2020/09; 2024-511083-90-00 (EU CTIS Number)
Record Dates: First submitted 2023-05-04; First posted 2023-05-15 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Wheezing; Wheezing Lower Respiratory Illness
Keywords: Innate immune response; Type 1 immune response; Type 2 immune response; Bacterial lysate; Immunomodulation; EAGLE
MeSH Terms: conditions — Respiratory Sounds

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OM-85 (Experimental): Patients will receive OM-85 capsules as a treatment for 6 months and will be under observation for 6 months.
  Interventions: Drug: OM-85
- Placebo (Placebo Comparator): Patients will receive placebo capsules as a treatment for 6 months and will be under observation for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OM-85 — OM-85 capsule (3.5mg) contents will be mixed with adequate quantity of water, fruit juice or milk/formula and orally administered once a day for 6 consecutive months.
  Arms: OM-85
Drug: Placebo — Placebo capsule contents will be mixed with adequate quantity of water, fruit juice or milk/formula and orally administered once a day for 6 consecutive months.
  Arms: Placebo

SUMMARY:
This study will assess the efficacy and safety of daily OM-85 treatment compared to placebo in children aged 6 months to 5 years with recurrent wheezing

DETAILED DESCRIPTION:
This study is a 12-months phase 2, randomized, double-blind, placebo-controlled, multicenter study to assess the efficacy and safety of daily treatment with OM-85 compared to placebo, when given on top of standard of care treatment, in reducing wheezing/asthma like episodes (WEs) during the 6-month treatment period in children aged 6 months to 5 years with previous recurrent WEs.

Patients will be randomized in a 1:1 ratio to OM-85 or placebo. The study consists of screening period (Day -20 to Day -1), a treatment period of 6 months, and an observational period of 6 months without treatment. Thus, the total duration of the study for each patient will be 12 months (±10 days) + up to 20 days for screening.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all the following criteria will be included in the study:

* Children of either gender, aged between 6 and 72 months (5 years inclusive).
* Children with recurrent wheezing:

  * For ICS/LTRA naïve patients or intermittent users (patients using ICS treatment only during an upper RTI to prevent WE): ≥2 WEs including at least 1 severe episode (i.e., treated with OCS OR having triggered an ED visit/hospitalization), OR ≥3 WEs including at least one that triggered an unscheduled physician visit, in the 12 months prior to enrollment.
  * For ICS/LTRA daily users: ≥1 severe WE (i.e., treated with OCS OR having triggered an ED visit/hospitalization) OR ≥2 WEs including at least one that triggered an unscheduled physician visit, as reported by parents or LAR of subject (i.e., guardians), in the 12 months prior to enrollment, while being on their daily controller therapy (at current dose or higher).
* Up-to-date vaccination status as per applicable State or country Vaccination Requirements for school/day-care entry.
* Parents or LAR have provided the appropriate written informed consent. Written informed consent must be provided before any study-specific procedures are performed including screening procedures.

Note: If a subject is experiencing respiratory symptoms at time of screening, he/she could only be randomized once symptoms have resolved for at least one week.

Exclusion Criteria:

* Known anatomic alterations of the respiratory tract.
* Wheezing documented to be caused by gastroesophageal reflux.
* Other known chronic respiratory diseases (e.g., tuberculosis or cystic fibrosis).
* Any known autoimmune disease.
* Known human immunodeficiency virus (HIV) infection or any known type of congenital or iatrogenic immune deficiency (including immunoglobulin (Ig) A deficiency).
* Known acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal function abnormalities.
* Children born prematurely i.e., before 34 weeks of gestational age.
* Children with an abnormally low or high weight for their age and height, if this would not allow safe completion of the clinical study in the opinion of the investigator.
* Any known neoplasia or malignancy.
* Treatment with the following medications:

  * Systemic corticosteroids within 4 weeks before study enrollment.
  * Previous and/or concomitant immunosuppressants, immunostimulants, or gamma globulins within 6 months before study enrollment.
* Any major surgery within the last 3 months prior to study enrollment or planned during the study duration.
* Known allergy or previous intolerance to investigational drug.
* Any other clinical conditions, which in the opinion of the Investigator, would not allow safe completion of the clinical study.
* Other household members have previously been randomized in this clinical study and have not completed their 6-month treatment period.
* Inability to comply with the study requested visit schedule (e.g., expected relocation within 12 months of the screening for the study).
* Currently enrolled in or has completed any other investigational device or drug study <30 days prior to screening or receiving other investigational agent(s).

Note: Subjects with past, present, or at risk of COVID-19 should not be excluded from the study.

Ages: 6 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 296 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Wheezing/Asthma like episodes (WEs) | 6 Months
  To assess the efficacy of OM-85 in reducing the rate of WEs compared to placebo during the 6-month Treatment period in children aged 6 months to 5 years with previous recurrent WEs.

SECONDARY OUTCOMES:
Rate of severe WEs | 6 Months
  To assess the efficacy of OM-85 in reducing the rate of severe WEs compared to placebo during the 6-month Treatment period.
Number of WE requiring oral corticosteroid (OCS) treatment during 6-month treatment period | 6 Months
  To assess the efficacy of OM-85 in reducing the use of oral corticosteroids for WEs compared to placebo during the 6-month Treatment period.
Number of days with WEs | 6 Months
  To assess the efficacy of OM-85 to decrease the cumulative number of days with WEs compared to placebo during the 6-month Treatment period.
Rate of WEs and severe WEs | From Month 6 up to Month 12
  To assess the efficacy of OM-85 compared to placebo in reducing the rate of WEs and severe WEs during the 6-month Observational period.
Number of WE requiring OCS treatments during 6-month observational period | From Month 6 up to Month 12
  To assess the efficacy of OM-85 in reducing the use of oral corticosteroids for WEs vs. placebo during the 6-month observational period.
Duration in days of WEs and severe WEs | 12 Months
  To assess the efficacy of OM-85 compared to placebo in reducing the duration of WEs and of severe WEs during the 6-month Treatment period and the 6-month Observational period.
Time to treatment failure | 12 Months
  To assess the efficacy of OM-85 compared to placebo to prolong time to treatment failure, during the whole study period.
Time to first, second and third WE | 12 Months
  To assess the efficacy of OM-85 compared to placebo to prolong the time to first, second, and third WE.
Number of routine asthma treatment | 12 Months
  To assess the efficacy of OM-85 compared to placebo to reduce the amount of routine asthma treatment required to control acute WEs during the 6-month treatment period and the 6-month observational period. The number of routine asthma treatment will be assessed.
Duration of routine asthma treatment | 12 Months
  To assess the efficacy of OM-85 compared to placebo to reduce the amount of routine asthma treatment required to control acute WEs during the 6-month treatment period and the 6-month observational period. The duration of routine asthma treatment will be assessed.
Percentage of patients with recurrent wheezing | 12 Months
  To assess the efficacy of OM-85 compared to placebo in reducing the percentage of patients with ≥1 WEs and ≥2 WEs during the 6-month treatment period and the 6-month observational period.
Number of days with respiratory tract infection (RTIs) symptoms | 12 Months
  To assess the efficacy of OM-85 compared to placebo in reducing the number of days with RTI symptoms during the 6-month treatment period and the 6-month observational period.
Level of severity of RTI symptoms (Absent/Mild/Moderate/Severe) | 12 Months
  To assess the efficacy of OM-85 compared to placebo in reducing the severity of RTI symptoms during the 6-month treatment period and the 6-month observational period. RTI symptoms severity will be assessed based on the symptom evaluation in the adapted Wisconsin Upper Respiratory Symptom Survey for Kids (WURSS-K), other relevant symptoms indicative of an RTI (e.g., headache, body aches), and tympanic temperature as recorded by patient's parents or legally authorized representative (LAR). Severity of symptoms will be determined by using the following definitions: child does not have this = absent (no sign/symptom evident); a little bad = mild (sign/symptom clearly present but easily tolerated); bad = moderate (definite awareness of sign/symptom that is bothersome but tolerable); and very bad = severe (sign/symptom that is hard to tolerate and causes interference with activities of daily life and/or sleeping).
Number of antibiotic cycles | 12 Months
  To assess the efficacy of OM-85 compared to placebo in reducing the antibiotics treatment for an RTI during the 6-month treatment period and the 6-month observational period.
Number of medical visits | 12 Months
  To assess the efficacy of OM-85 compared to placebo in reducing the number of medical visits (hospitalizations, visits to emergency rooms, or to a physician/health care provider) due to respiratory events during the 6-month treatment period and the 6-month observational period.
Number of days absent from daycare/school | 12 Months
  To assess the efficacy of OM-85 compared to placebo in reducing the number of days of absence from daycare/school due to respiratory events during the 6-month treatment period and the 6-month observational period.
Number of patients with adverse events (AEs) | 12 Months
  To assess the safety of daily OM-85 treatment compared to placebo in children aged 6 months to 5 years with recurrent WEs during the 6-month treatment period and the 6-month observational period.
Number of work days when parents/LAR had to miss work or had their productivity | 12 Months
  To assess the efficacy of OM-85 compared to placebo in reducing the number of days of absence from daycare/school due to respiratory events during the 6-month treatment period and the 6-month observational period.

CONTACTS AND LOCATIONS:
Locations (37):
- United States (30):
  - Arizona Medical Clinic, Phoenix, Arizona
  - Phoenix Children's Hospital, Phoenix, Arizona
  - The University of Arizona Medical Center - University Campus, Tucson, Arizona
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Kern Research Inc., Bakersfield, California
  - Hoag Health Center Foothill Ranch, Foothill Ranch, California
  - UCSF Benioff Children's Hospital Oakland Primary Care Clinic, Oakland, California
  - Allergy & Asthma Medical Group and Research (AAMGRC) - Allergy, Asthma and Immunology, San Diego, California
  - Rady Children's Hospital, San Diego, California
  - Children's Hospital Colorado - Pediatric Heart Lung Center - Pediatrics, Aurora, Colorado
  - BioMD Clinical Research, Coral Gables, Florida
  - C & R Research Services USA. Inc, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Riley Children's Health - Pediatrics, Indianapolis, Indiana
  - Allergy & Asthma Specialists PSC, Owensboro, Kentucky
  - Velocity Clinical Research - Lafayette, Lafayette, Louisiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Velocity Clinical Research - Binghamton, Binghamton, New York
  - Northwell Health/Division of Allergy & Immunology, Great Neck, New York
  - UNC Hospitals, The Univ of NC at Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children'S Hospital Medical Center, Cincinnati, Ohio
  - Allergy, Asthma and Clinical Research Center, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - Monroe Carell Jr. Children's Hospital, Nashville, Tennessee
  - Helios Clinical Research - Houston, Houston, Texas
  - La Providence Pediatrics Clinic, Houston, Texas
  - Prime Clinical Research Inc, Mansfield, Texas
  - STAAMP Research, San Antonio, Texas
  - The University of Texas Health Science Center at Tyler - Pulmonology, Tyler, Texas
  - University of Wisconsin School of Medicine & Public Health - allergy, Pulmonary, & Critical Care Medicine, Madison, Wisconsin
- Australia (2):
  - University Hospital Geelong - Barwon Health, Geelong, Victoria
  - The Royal Childrens Hospital, Melbourne, Victoria
- Hungary (2):
  - Borsod-Abauj-Zemplen Varmegyei Kozponti Korhaz, Miskolc, Borsod-Abauj Zemplen county
  - Aranyklinika Kft., Szeged, Csongrád megye
- Poland (3):
  - ALERGO-MED Specjalistyczna Przychodnia Lekarska Sp.z o. o., Tarnów, Lesser Poland Voivodeship
  - NZOZ E-Vita, Bialystok, Podlaskie Voivodeship
  - Velocity Skierniewice Sp. z o.o., Skierniewice, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: No